CLINICAL TRIAL: NCT03235752
Title: A Phase II, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Safety and Efficacy of TJ301 (FE 999301) Administered Intravenously in Patients With Active Ulcerative Colitis
Brief Title: Safety and Efficacy of TJ301 IV in Participants With Active Ulcerative Colitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: I-Mab Biopharma HongKong Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CTJ301UC201
Record Dates: First submitted 2017-07-28; First posted 2017-08-01 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2020-12

CONDITIONS: Active Ulcerative Colitis
Keywords: Randomized; Double-blind; Placebo-controlled; Safety; Efficacy; Active Ulcerative Colitis

STUDY DESIGN:
Intervention Model Description: Randomized, Double-blind, Placebo-controlled
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Randomized, Double-blind, Placebo-controlled
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- TJ301 300mg (Experimental): TJ301 300mg administrations will occur on Days 0, 14, 28, 42, 56, and 70.
  Interventions: Drug: TJ301 300mg
- TJ301 600mg (Experimental): TJ301 300mg administrations will occur on Days 0, 14, 28, 42, 56, and 70.
  Interventions: Drug: TJ301 600mg
- Placebo (Placebo Comparator): Placebo administrations will occur on Days 0, 14, 28, 42, 56, and 70.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TJ301 300mg — TJ301 300mg IV infusion
  Arms: TJ301 300mg
Drug: TJ301 600mg — TJ301 600mg IV infusion
  Arms: TJ301 600mg
Drug: Placebo — Placebo IV infusion
  Arms: Placebo

SUMMARY:
This is a multicenter, randomized, double-blind, placebo-controlled phase II study.

DETAILED DESCRIPTION:
is a multicenter, randomized, double-blind, placebo-controlled phase II study. The trial includes a Run-in Period (if stable conventional treatment needed), a 4-week Screening Period, a 12-week Treatment Period, and a 3-week Safety Follow-up Period to Day 105.

90 patients will be centrally, dynamically, randomly assigned to 3 groups (1:1:1) to receive 600mg TJ301 Q2W, 300mg TJ301 Q2W or placebo Q2W.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients 18-70 (inclusive) years of age.
2. Hisory of active UC of more than 3 months. Active UC confirmed by colonoscopy with biopsy or flexible sigmoidoscopy with biopsy at Screening, with extending > 15-cm past the anal verge from endoscopy. Biopsy sample is not necessary if UC is already confirmed.
3. Active UC with a full Mayo score≥5 and a rectal bleeding subscore ≥1 at screening.
4. During Day -28 to Day -6 prior to Randomisation, an endoscopy subscore ≥2.
5. Treated with conventional non-biological UC therapy: with corticosteroids stable for at least 2 weeks prior to Randomization at no more than 20 mg prednisone per day (or equivalent), and/or with medications containing 5-aminosalicylates (5-ASA) at no less than 2 g 5-ASA per day for at least 3 months and stable for at least 4 weeks prior to Randomization, and/or with azathioprine (AZA) at no less than 0.75 mg/kg/day or mercaptopurine (6-MP) at no less than 0.5 mg/kg/day for at least 6 months and stable for at least 6 weeks prior to Randomization, or MTX no less than 12.5 mg/week and stable for at least 12 weeks prior to Randomization.
6. Male subjects and female subjects of child bearing potential must have been willing to practice effective contraception during the study and been willing and able to continue contraception for 1 month after their last dose of the study treatment.
7. The patient is able and willing to comply with the requirements of this trial protocol.
8. The subject should be able to read and write to understand and fill out Patient Diary.
9. Voluntarily signed Informed Consent obtained before any trial-related procedures are performed.
10. The subject have not received any biologic therapies OR have received 1 biologic drug for the treatment of UC or immune diseases and the last dose must be longer than 8-week or a 5 half-life (whichever is longer) period prior to the first dose of study drug.

Exclusion Criteria:

1. Pregnant or breastfeeding women.
2. Contraindication to colonoscopy or sigmoidoscopy.
3. Allergies to any component of TJ301.
4. Subject who is likely to receive surgery for UC treatment within 1 month based on investigator's evaluation.
5. History of colostomy, colectomy or partial colectomy.
6. Current diagnosis of inflammatory bowel disease unclassified, Crohn's disease, ischemic colitis, fulminant colitis and/or toxic megacolon, patients with ulcerative colitis limited to the rectum (ulcerative proctitis), infective enteritis, amebic bowel disease or intestinal schistosomiasis.
7. History of malignancy other than a successfully treated non-metastatic cutaneous squamous cell or basal cell carcinoma and/or localized carcinoma in situ of the cervix. If the Screening colonoscopy shows evidence of dysplasia or a malignancy, the patient is not eligible.
8. Primary or secondary immunodeficiency including neutropenia (absolute neutrophil count <1500/μL); or lymphopenia (absolute lymphocyte count <500/μL).
9. Moderate to severe anaemia (haemoglobin <9 g/dL), or thrombocytopenia (platelet count <75 000/μL), or serum creatinine >2 mg/dL.
10. Autoimmune disease besides UC, with the exceptions of Sjogren's syndrome or hypothyroidism.
11. Clostridium (C.) difficile positive at screening visit or treated for C. difficile within the 4 weeks prior to Randomization.
12. serum transaminases >2.5 x upper limit of normal [ULN], alkaline phosphatase >2.5 x ULN.
13. Serious underlying disease other than UC in the opinion of the investigator.
14. History of drug addiction within the last 1 year or current drug addiction or use of illicit drugs.
15. Any indication of the regular use of more than 40 grams of alcohol every day.
16. Smokers who smoke more than 10 cigarettes per day.
17. Known concurrent acute or chronic viral hepatitis B or C infection or human immunodeficiency virus (HIV) infection.
18. Presence or history of active tuberculosis (TB) or latent TB infection, defined as 1) a positive QuantiFERON-TB Gold test at Screening; or 2) a T-spot test within 4 weeks of Randomisation and evidence of current or previous pulmonary tuberculosis by low-dose CT or chest X-ray within 12 weeks of Randomisation. Patients with old TB will also be excluded.
19. Positive immunoglobulin M antibody titres to Epstein-Barr virus (EBV).
20. Subjects with positive results for cytomegalovirus at screening are to be excluded.
21. Receiving any investigational therapy or any approved therapy for investigational use within 30 days or 5 half-lives prior to Randomization (whichever is longer).
22. Currently taking any medications other than those allowed per protocol guidelines.
23. Infections (including diverticulitis) requiring treatment with antibiotics, antivirals, or antifungals within 14 days prior to Randomisation.
24. Received any live (attenuated) vaccines within 30 days prior to Randomisation.
25. Recent treatment with medium-to-high-dose intravenous corticosteroids (methylprednisolone 60 mg/day or hydrocortisone 300 mg/day) within 8 weeks prior to Randomisation or oral corticosteroids of more than 20 mg prednisone per day (or equivalent).
26. Receipt of cyclosporine, tacrolimus, sirolimus, thalidomide, or mycophenolate mofetil within 30 days prior to Randomisation.
27. Treatment with therapeutic enema or suppository, other than required for endoscopy preparation, within 14 days prior to the screening endoscopy and during the remainder of the trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2018-02-06 (Actual); Primary Completion 2020-12-21 (Actual); Study Completion 2020-12-21 (Actual)

PRIMARY OUTCOMES:
Clinical and endoscopy response | Week 12
  Clinical and endoscopy response (decrease from Baseline in full Mayo score ≥3 and ≥30%, including decrease from Baseline in rectal bleeding subscore ≥1 or rectal bleeding subscore ≤1) at Week 12.

SECONDARY OUTCOMES:
Clinical and endoscopy remission at Week 12 | Week 12.
  Clinical and endoscopy remission at Week 12, defined as a full Mayo score ≤2, no individual subscore >1, rectal bleeding subscore = 0.
Clinical remission at Weeks 4, 6, 8, 10, and 12 | Weeks 4, 6, 8, 10, and 12
  Clinical remission at Weeks 4, 6, 8, 10, and 12 defined as a stool frequency subscore=0, rectal bleeding subscore = 0, and 9-point partial Mayo score ≤1.

OTHER OUTCOMES:
Change from Baseline to Weeks 4, 8, and 12 in exploratory biomarkers | Baseline to Weeks 4, 8, and 12
  Change from Baseline to Weeks 4, 8, and 12 in exploratory biomarkers (erythrocyte sedimentation rate [ESR], C-reactive protein (CRP), IL-6, IL-6/sIL-6R complex, neutrophil and platelet count, faecal calprotectin).

CONTACTS AND LOCATIONS:
Overall Officials: Minhu Chen, Doctor, Principal Investigator — First Affiliated Hospital, Sun Yat-Sen University
Locations (27):
- China (22):
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Beijing Friendship Hospital Affiliated to the Capital University of Medical Sciences, Beijing, Beijing Municipality
  - The Seventh Medical Center of PLA Army General Hospital, Beijing, Beijing Municipality
  - West China Hospital of Sichuan University, Sichuan, Chengdu
  - The Sixth Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangzhou
  - Guangdong Provincial People's Hospital, Guangzhou, Guangzhou
  - Nanfang Hospital of SMU, Guangzhou, Guangzhou
  - The First Affiliated Hospital, Sun Yat-sen University, Guanzhou, Guangzhou
  - Hainan General Hospital, Hainan, Hainan
  - Sir Run Run Shaw Hospital Zhejiang University, School of Medicine, Zhejiang, Hangzhou
  - The First Affiliated Hospital of Harbin Medical University, Harbin, Harbin
  - The first Bethune hospital of Jilin university, Jilin, Jilin
  - The first affiliated hospital of Nanchang Univesity, Nanchang, Nanchang
  - Jiangsu Province Hospital, Nanjing, Nanjing
  - The Affiliated Hospital of Nanjing University Medical School, Nanjing, Nanjing
  - Zhongda Hospital Southeast University, Nanjing, Nanjing
  - Renji Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality
  - Ruijin Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality
  - Xin Hua Hospital affiliated to Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality
  - Shengjing hospital of China medical university, Shenyang, Shenyang
  - Second Hospital of Shanxi Medical University, Shanxi, Taiyuan
  - Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality
- South Korea (2):
  - Yeungnam University Medical Center, Daegu
  - CHA Bundang Medical Center, CHA University, Seoul
- Taiwan (3):
  - National Taiwan University Hospital, Kaohsiung City
  - Chang Gung Memorial Hospital, Taipei
  - Chang Gung Memorial Hospital, Taoyuan District

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhang S, Chen B, Wang B, Chen H, Li Y, Cao Q, Zhong J, Shieh MJ, Ran Z, Tang T, Yang M, Xu B, Wang Q, Liu Y, Ma L, Wang X, Zhang N, Zhang S, Guo W, Huang L, Schreiber S, Chen M. Effect of Induction Therapy With Olamkicept vs Placebo on Clinical Response in Patients With Active Ulcerative Colitis: A Randomized Clinical Trial. JAMA. 2023 Mar 7;329(9):725-734. doi: 10.1001/jama.2023.1084. PMID 36881032